CLINICAL TRIAL: NCT04169113
Title: How Many Opiates Should be Prescribed for Pain in Patients Undergoing Hip Arthroscopy?
Brief Title: Opiate Prescribing Guidelines Following Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Vehniah Tjong, Assistant Professor of Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00207356
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Hip Injuries
Keywords: Hip Arthroscopy; Opiate Use
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Hip Arthroscopy (Active Comparator): Will be prescribed 60 opiate tablets in addition to other routine post-operative pain medication regimens.
  Interventions: Other: Group 1 - Opiate Tablets post Hip Arthroscopy
- Group 2 - Hip Arthroscopy (Active Comparator): Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
  Interventions: Other: Group 2 - Opiate Tablets post Hip Arthroscopy

INTERVENTIONS:
Other: Group 1 - Opiate Tablets post Hip Arthroscopy — Will be prescribed 60 opiate tablets in addition to other routine post-operative pain medication regimens.
  Arms: Group 1 - Hip Arthroscopy
Other: Group 2 - Opiate Tablets post Hip Arthroscopy — Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
  Arms: Group 2 - Hip Arthroscopy

SUMMARY:
The purpose of the study is to determine if opiates are required to achieve appropriate analgesia after hip arthroscopy in outpatient surgery. The investigators hypothesize that patients are frequently prescribed more opiates than are needed after surgery, resulting in excess medications that are at risk for misuse, diversion and contribution to the opioid epidemic

DETAILED DESCRIPTION:
Perioperative pain management is an important aspect of quality patient care. Opioid pain medications are increasingly being used for pain control, with the United States writing over 250 million prescriptions for painkillers per year. Increased usage has led to unintended negative consequences for individuals and society. It is estimated that 46 people die each day from an overdose of prescription painkillers, and individual use can lead to the development of tolerance and worse treatment outcomes. Further issues arise when opioids are misused, it is estimated that nontherapeutic use has increased three fold in recent years. In the United States alone in 2006 the estimated total cost of opioid prescription misuse was $53.4 billion, of which $42 billion was attributed to lost productivity, $8.2 billion to criminal justice cost and the remainder drug abuse treatment and medical complications. The federal government has recognized this epidemic and raised a call for clinicians to more responsibly prescribe opiate pain medications

Opiate use has increased in recent years, from 2000-2010 the use of opiates in office based visits nearly doubled from 11.3% to 19.6% whereas there was no change in the prescribing of non-opioid pharmacotherapies. Further, when specifically looking at new musculoskeletal pain visits, one half resulted in pharmacologic treatment, with the prescribing of non-opioid pharmacotherapies decreasing from 38% to 29% from 2000 to 2010, respectively. The clinical use of opioids for post-operative pain control has also been linked to the opioid epidemic and risk of future abuse. Legitimate opioid use before high school graduation is independently associated with a 33% increased risk of future misuse after high school.

It has been estimated that orthopedic surgeons prescribe 7.7% of all opioids in the United States.Special attention needs to be paid to the amount of opioid pain medications orthopedic surgeons prescribe to patients after ambulatory surgery, there is considerable variability among surgeon and procedure in regards to the amount of opioids to prescribe with many patients left with excess unused medication .An analysis of 250 patients undergoing outpatient upper extremity surgery found that on average patients consumed 10 opioid pills, with 19 pills left over and a total of 4,639 pills going unused in the cohort. Leftover prescription opioids are at risk for diversion to family and friends for nonmedical use. Further studies are needed to quantify the amount of opioids to prescribe for specific orthopedic procedures to limit excess narcotic use, misuse, diversion and contribution to the opioid epidemic.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Northwestern Memorial Hospital (NMH) or to a Northwestern orthopaedic surgery faculty member's clinic undergoing hip arthroscopy
* 18 years old or greater
* Ability to read and speak English

Exclusion Criteria:

* Revision surgery
* Oncologic etiology
* Arthroscopic hip surgery that involves procedures other than labral repair, acetabuloplasty, CAM-plasty, IT band windowing, Iliopsoas lengthening
* Patients with a current indication of narcotic use
* Individuals unable to provide informed consent:
* Prisoners
* Pregnant women
* Minors/Individuals under 18 years of age

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Department of Orthopaedic Surgery, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (60) - Hip Arthroscopy: Will be prescribed 60 opiate tablets in addition to other routine post-operative pain medication regimens.
  Group 1 - Opiate Tablets post Hip Arthroscopy: Will be prescribed 60 opiate tablets in addition to other routine post-operative pain medication regimens.
- Group 2 (30) - Hip Arthroscopy: Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
  Group 2 - Opiate Tablets post Hip Arthroscopy: Will be prescribed 30 opiate tablets in addition to other routine post-operative pain medication regimens.
Period: Overall Study
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Started | 52 | 59
Completed | 47 | 53
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Hip Arthroscopy | Group 2 - Hip Arthroscopy | Total
Number analyzed (Participants) | 52 | 59 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 59 | 111
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (11.2) | 36.9 (11.8) | 37.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 73
  Male | 14 | 24 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Are you an active smoker? [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 4
  No | 50 | 57 | 107
If no, have you ever consistently smoked cigarettes (daily for > 1 month)? [Count of Participants; unit: Participants]
  Yes | 6 | 10 | 16
  No | 46 | 49 | 95
What is your employment status? [Count of Participants; unit: Participants]
  Employed | 39 | 48 | 87
  Unemployed | 11 | 11 | 22
  Disabled | 2 | 0 | 2
Is this injury part of a workers compensation claim? [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 2
  No | 51 | 58 | 109
Are you currently using narcotic pain medications (ex. Norco, Vicodin, Oxycontin/codone)? [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 51 | 59 | 110
Do you have a personal history of illicit substance abuse? [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 51 | 59 | 110
Do you have a family history of substance abuse (ex. prescription or illicit drugs, alcohol)? [Count of Participants; unit: Participants]
  Yes | 9 | 8 | 17
  No | 43 | 51 | 94
What is the highest level of education you attained? [Count of Participants; unit: Participants]
  Completed High School | 5 | 12 | 17
  Undergraduate | 31 | 30 | 61
  Graduate | 16 | 17 | 33
What is your average yearly household income? [Count of Participants; unit: Participants]
  Less than $20,000 | 4 | 3 | 7
  $20,000 -$34,999 | 1 | 3 | 4
  $35,000 -$49,999 | 4 | 5 | 9
  $50,000 -$74,999 | 5 | 8 | 13
  $75,000 - $99,999 | 8 | 10 | 18
  $100,000 -$149,999 | 11 | 8 | 19
  $150,000 - $199,999 | 6 | 10 | 16
  $200,000 or more | 12 | 12 | 24
  missing | 1 | 0 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.2 (5.5) | 27.8 (6.1) | 27.1 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Scores
Description: minimum score: 0 = no pain, maximum score: 10 = worst imaginable pain; lower value indicates less pain reported by the patient
Time Frame: Baseline (pre-operative)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 52 | 59
score on a scale | 4.2 (2.6) | 4.0 (1.7)

2. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Scores
Description: as for outcome 1
Time Frame: 2 hours post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
score on a scale | 5.0 (2.1) | 4.7 (2.1)

3. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Scores
Description: as for outcome 1
Time Frame: 24 hours post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
score on a scale | 3.9 (2.5) | 3.8 (2.3)

4. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Scores
Description: as for outcome 1
Time Frame: 48 hours post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
score on a scale | 3.2 (2.4) | 3.3 (2.1)

5. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Scores
Description: as for outcome 1
Time Frame: 7 days post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
score on a scale | 2.3 (2.4) | 2.2 (1.6)

6. Primary Outcome: Opiates Taken
Description: Number of prescribed narcotic pills taken in the preceding time period
Time Frame: 24 hours post-operative
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
tablets | 3.0 (2.2) | 2.4 (2.5)

7. Primary Outcome: Opiates Taken
Description: Number of prescribed narcotic medication tablets taken in the preceding time period
Time Frame: 48 hours post-operative
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
tablets | 5.2 (5.7) | 4.9 (5.9)

8. Primary Outcome: Opiates Taken
Description: Number of prescribed narcotic medication tablets taken in the preceding time period
Time Frame: 7 days post-operative
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
tablets | 10.4 (15.9) | 8.8 (9.3)

9. Primary Outcome: Opiates Taken
Description: Number of prescribed narcotic medication tablets taken in the preceding time period
Time Frame: 21 days post-operative
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
tablets | 10.5 (16.5) | 9.2 (11.1)

10. Primary Outcome: Opiates Remaining
Description: Number of prescribed narcotic medication tablets remaining from initial amount prescribed
Time Frame: 24 hours post-operative
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
tablets | 57.0 (2.2) | 27.6 (2.5)

11. Primary Outcome: Opiates Remaining
Description: Number of prescribed narcotic medication tablets remaining from initial amount prescribed
Time Frame: 48 hours post-operative
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
tablets | 54.8 (5.7) | 25.1 (5.9)

12. Primary Outcome: Opiates Remaining
Description: Number of prescribed narcotic medication tablets remaining from initial amount prescribed
Time Frame: 7 days post-operative
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
tablets | 49.6 (15.9) | 22.3 (8.4)

13. Primary Outcome: Opiates Remaining
Description: Number of prescribed narcotic medication tablets remaining from initial amount prescribed
Time Frame: 21 days post-operative
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
tablets | 49.5 (16.5) | 22.0 (7.9)

14. Primary Outcome: Date of Last Opiate Taken
Description: Days following surgery that the most recent dose of narcotic medication was taken
Time Frame: 21 days post-operative
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
days | 5.0 (4.9) | 4.6 (5.8)

15. Primary Outcome: Numeric Pain Rating Scale (NPRS) Pain Scores
Description: as for outcome 1
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
score on a scale | 2.6 (2.3) | 2.0 (1.8)

16. Primary Outcome: Number of Participants Reporting Side Effects
Description: As reported by patient. Including: blurred vision, confusion/mental fog, constipation, dizziness, drowsiness, itchiness, nausea/vomiting
Time Frame: 24 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
Participants
  Yes | 16 | 18
  No | 31 | 35

17. Primary Outcome: Number of Participants Reporting Side Effects
Description: As reported by patient. Including: blurred vision, confusion/mental fog, constipation, dizziness, drowsiness, nausea/vomiting
Time Frame: 48 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
Participants
  Yes | 15 | 14
  No | 32 | 39

18. Primary Outcome: Number of Participants Reporting Side Effects
Description: as for outcome 17
Time Frame: 7 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
Participants
  Yes | 10 | 8
  No | 37 | 45

19. Primary Outcome: Number of Participants Reporting Side Effects
Description: as for outcome 17
Time Frame: 21 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
Number analyzed (Participants) | 47 | 53
Participants
  Yes | 9 | 7
  No | 38 | 46

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Group 1 (60) - Hip Arthroscopy | Group 2 (30) - Hip Arthroscopy
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/59
Other Adverse Events (participants affected / at risk) | 0/52 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT04169113/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04169113/SAP_001.pdf